CLINICAL TRIAL: NCT03376568
Title: Feature of Polysomnography and Cerebral Metabolism and Function in Narcolepsy With/Without RBD and Control Subject
Brief Title: Investigation of Clinical Feature and Brain Function in Narcoleptic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDLL-201601-08
Record Dates: First submitted 2017-12-04; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Narcolepsy; REM Sleep Behavior Disorder
Keywords: polysomnographic; multiple sleep latency test; fMRI
MeSH Terms: conditions — Narcolepsy; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Narcolepsy with RBD & Control: Narcolepsy with REM sleep disorder lable(20) and Control subjects lable(20)
- Narcolepsy with /without RBD: Narcolepsy with REM sleep disorder lable(20) and Narcolepsy without REM sleep disorderlable (20)

SUMMARY:
This study evaluates the PSG and cerebral metabolism and functions in narcolepsy with/without RBD

DETAILED DESCRIPTION:
Polysomnographic (PSG) work-up one night to record nocturnal sleep condition in narcolepsy with /without RBD and control subjects including sleep macrostructure, occurrence of sleep onset rapid eye movement period(SOREMP), sleep stages distribution, and sleep arousle and leg movement and apnea hyponea index would be calculated.

Functional magnetic resonance imaging (fMRI) has been used in human to nonivasiverlyn investigate the neural mechanisms. This technique also apply to measures the variations in brain perfusion, structure and morphology in narcolepsy patients by assessing the blood oxygen level-dependent (BOLD) signal diffusion tensor imaging (DTI and voxel-based morphometry(VBM)

This study compare the feature of PSG and fMRI between narcolepsy with RBD, narcolepsy without RBD, control subject to evaluates the PSG and cerebral metabolism and functions in narcolepsy with/without RBD.

ELIGIBILITY:
Inclusion Criteria:

* Narcolepsy meet to the international classification of sleep disorder,3rd edition (ICSD-3) , and RBD meet to the minimal diagnostic criteria according to the international Classification of Sleep, control subjects .

Exclusion Criteria:

History of heart disease History of central nervous system organic psychosis AHI>15次/h History of alcohol dependence and drug abuse

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will need about 40 narcoleptic patients with /without RBD between 10 and 65 years of age,and about 20 age- and gender-matched control subjects.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
video-polysomnographic(PSG) | up to 100 weeks
  video-PSG monitor sleep from 9:00pm to 6:00am

SECONDARY OUTCOMES:
multiple sleep latency test (MSLT) | up to 100 weeks
  MSLT in the next day of PSG record daytime sleepiness
functional magnetic resonance imaging (fMRI) | up to 100 weeks
  All narcolepsy with or withoutRBD accepts fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China